CLINICAL TRIAL: NCT03485599
Title: Prevalence,Knowledge and Attitude of HIV /AIDS in Luxor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zienab Gamea, Principal Investigator, Assiut University
Other Study IDs: PKHIVL
Record Dates: First submitted 2018-03-21; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV infected people: Blood samples will be taken and rapid HIV test by ELIZA will be done ,for positive cases Westron blot done
  Interventions: Diagnostic Test: ELIZA , Westron blot

INTERVENTIONS:
Diagnostic Test: ELIZA , Westron blot — Blood sample will be taken then rapid test by ELIZA will be done if positive then confirmatory test by Westron blot will be done

SUMMARY:
Human immunodeficiency virus infection is a global pandemic problem. About 35.3 million infected people in the world, so causing a great social, economical, political and cultural problems worldwide.

In 1986 Egypt's first AIDS case was discovered , since then the number of infected cases cases are increasing.According to United Nations 2016 statistics, there are about 11,000 infected people living with Human immunodeficiency virus in Egypt.

DETAILED DESCRIPTION:
Human immunodeficiency virus is a lentivirus that causes the infection and over time leading to Acquired immunodeficiency syndrome.

The virus spread primarily by unprotected sex including vaginal, anal and oral sex, contaminated blood transfusions, infected needles, and from mother to child during pregnancy, delivery, or from milk during breastfeeding.

In 1986 Egypt's first AIDS case was discovered , since then the number of infected cases cases are increasing.According to United Nations 2016 statistics, there are about 11,000 infected people living with Human immunodeficiency virus in Egypt.

According to the National Aids Program, the primary mode of transmission is heterosexual intercourse, followed by homosexual intercourse , renal dialysis , and blood transfusion Others include street children, prisoners, and refugees, female sex workers, men have sex with men, and injecting drug users.

Human immunodeficiency virus related stigma and discrimination is a great barrier to effectively fighting the disease epidemic.

This study will assess prevalence, knowledge, attitudes of Human immunodeficiency virus and Acquired immunodeficiency syndrome people in Luxor Governorate in Upper Egypt.

ELIGIBILITY:
Inclusion Criteria:

1-People living in Luxor. 2 Subjects of high risk groups as men have sex with men, children street, female sex workers.

3-People clinically diagnosed as HIV/AIDS. 4-People in contact with HIV/AIDS patients.

Exclusion Criteria:

1 - Subjects outside Luxor 2- People refused to consent 3- Mentally disordered patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community based cross sectional study will be done in Luxor,Data will be collected by physicians at the mobile Voluntary Confidential Counseling and Testing centers apart of National strategic plan , blood samples will be taken by laboratory technician,diagnostic tests will be done.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
knowledge score | 20 mintues
  Questionnaire to define knowledge score of HIV/AIDS through an interview

CONTACTS AND LOCATIONS:
Overall Officials: Hisham Zayan, Assistant, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cohen MS, Hellmann N, Levy JA, DeCock K, Lange J. The spread, treatment, and prevention of HIV-1: evolution of a global pandemic. J Clin Invest. 2008 Apr;118(4):1244-54. doi: 10.1172/JCI34706. PMID 18382737
- [Result] Abstracts from the 38th annual meeting of the society of general internal medicine. J Gen Intern Med. 2015 Apr;30 Suppl 2(Suppl 2):45-551. doi: 10.1007/s11606-015-3271-0. No abstract available. PMID 25869016
- [Result] Getnet MK, Damen HM. Level of stigma among female sex workers: comparison of two surveys of HIV behavioral data, Ethiopia. Afr Health Sci. 2011 Dec;11(4):543-9. PMID 22649433